CLINICAL TRIAL: NCT00586066
Title: Memantine and Cognitive Dysfunction in Bipolar Disorder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Forest Laboratories (Industry)
Responsible Party: Principal Investigator, Andrew A. Nierenberg, MD, Director, Bipolar Clinic and Research Program, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2005-p-001651; NCT00645476 (obsolete NCT alias)
Record Dates: First submitted 2007-12-21; First posted 2008-01-04 (Estimated); Results first posted 2017-05-05 (Actual); Last update posted 2017-10-06 (Actual); Status verified 2017-09

CONDITIONS: Bipolar Disorder
Keywords: Bipolar disorder; Cognitive dysfunction; Memantine; NMDA antagonist
MeSH Terms: conditions — Bipolar Disorder; Cognitive Dysfunction | interventions — Memantine; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Placebo-matching memantine 5 mg tablet once per day for 1 week; dose increase if tolerated to placebo-matching memantine 5 mg twice a day, in the morning and the evening in Week 2; dose increase if tolerated to placebo-matching memantine 5 mg in the morning and placebo-matching memantine 10 mg in the evening in Week 3; dose increase if tolerated to placebo-matching memantine 10 mg twice a day, in the morning and the evening Weeks 4 to 12.
  Interventions: Drug: Placebo
- Memantine (Experimental): Re-purposed Alzheimer's drug to treat cognitive dysfunction associated with bipolar disorder. Memantine 5 mg tablet once per day for 1 week; dose increase if tolerated to memantine 5 mg twice a day, in the morning and the evening in Week 2; dose increase if tolerated to memantine 5 mg in the morning and memantine 10 mg in the evening in Week 3; dose increase if tolerated to memantine 10 mg twice a day, in the morning and the evening Weeks 4 to 12.
  Interventions: Drug: Memantine

INTERVENTIONS:
Drug: Memantine — Week 0: 5 mg memantine or placebo once a day (q.d.) Week 1: 5 mg memantine or placebo twice a day (b.i.d.) Week 2-3: 5 mg memantine or placebo once in the morning (q.a.m.)/10 mg once in the evening (q.p.m.) Week 4-12: 10mg Memantine or placebo b.i.d.
  Other Names: Namenda
  Arms: Memantine
Drug: Placebo — Inactive comparator. Placebo-matching memantine tablet.
  Other Names: Sugar pill
  Arms: Placebo

SUMMARY:
The purpose of this study is to see whether memantine improves memory function in participants with bipolar disorder who have minimal symptoms. Secondary analyses will test the role of memantine in improving residual mood symptoms (depression and mania) in participants with bipolar disorder.

We hypothesize that in participants with bipolar disorder who have minimal symptoms memantine will be effective in improving cognitive functions, as measured by the difference in neuropsychological test scores at the beginning and at the end of the trial.

DETAILED DESCRIPTION:
A large proportion of participants with bipolar disorder experience significant cognitive dysfunction, even when euthymic, after adequate treatment. The cognitive deficits in asymptomatic patients with bipolar disorder are very important for the participant's psychosocial function. In this population, cognitive deficits have been associated with poor psychosocial functioning, such as inability to hold a job. Memantine is a glutamate N-methyl-D-aspartate (NMDA) receptor antagonist which has shown efficacy in cognitive dysfunction due to moderate to severe Alzheimer disease.

Demonstrating the role of memantine in reducing cognitive dysfunction in minimally symptomatic participants with bipolar disorder promises to provide important clinical information, which could lead to improvements in well-being and functional status for large populations of participants with bipolar disorder.

ELIGIBILITY:
Inclusion Criteria:

* Diagnostic and Statistical Manual-IV (DSM-IV) diagnostic criteria for any bipolar disorder [type I, type II, and not otherwise specified (NOS)] (diagnosed with the use of the Structured Clinical Interview for DSM-IV-TR Mood Module (SCID Mood Module)
* Written informed consent
* Men or women aged 18-65
* A baseline Hamilton-D 17 score of < 10 at screen and baseline visits.
* A baseline Young Mania Rating Scale score of < 10 at screen and baseline visits.
* No acute episodes of depression or mania for the previous 12 weeks.
* Massachusetts General Hospital Cognitive and Physical Functioning Scale: Cut-off: >15 or Everyday Cognition Self-Report Form: Average of all items >1.5 or Repeatable Battery for the Assessment of Neuropsychological Status (RBANS): <12 years education, RBANS total scale score of <85 =12 years education, RBANS total scale score of <93 >12 years education, RBANS total scale score of <100
* Able to read and understand English.

Exclusion Criteria:

Patients meeting any of the following criteria will be excluded from the study:

* Participants with suicidal ideation where outpatient treatment is determined unsafe by the study clinician. These patients will be immediately referred to appropriate clinical treatment.
* Pregnant women, nursing mothers, or women of childbearing potential who are not using a medically accepted means of contraception (defined as oral contraceptive pill or implant, condom, diaphragm, spermicide, intrauterine device (IUD), s/p tubal ligation, partner with vasectomy).
* Serious or unstable medical illness, including liver impairment, kidney impairment, cardiovascular, hepatic, respiratory, endocrine, neurologic or hematologic disease.
* History of seizure disorder, brain injury, any history of known neurological disease [multiple sclerosis, degenerative disease such as amyotrophic lateral sclerosis (ALS), Parkinson disease and any movement disorders, etc].
* History or current diagnosis of the following DSM-IV psychiatric illness: organic mental disorder, schizophrenia, schizoaffective disorder, delusional disorder, psychotic disorders not otherwise specified, major depressive disorder, patients with substance dependence disorders, including alcohol, active within the last 12 months.
* History of multiple adverse drug reactions.
* Patients with mood congruent or mood incongruent psychotic features within the last 12 months.
* Clinical or laboratory evidence of hypothyroidism.
* Patients who have had an episode of acute depression or mania during the 12 weeks prior to enrollment.
* Patients who have had electroconvulsive therapy (ECT) within the 6 months preceding enrollment.
* Patients taking drugs which alkalinize the urine.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2005-11 (Actual); Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew A. Nierenberg, M.D., Principal Investigator — Massachusetts General Hospital
Locations (3):
- United States (3):
  - Cedars Sinai Department of Psychiatry, Los Angeles, California
  - Asher Depression Center, Northwestern University, Chicago, Illinois
  - Massachusetts General Hospital, Boston, Massachusetts

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment began in November 2005 and closed in December 2009.
Groups:
- Memantine: Memantine 5 mg tablet once per day for 1 week; dose increase if tolerated to memantine 5 mg twice a day, in the morning and the evening in Week 2; dose increase if tolerated to memantine 5 mg in the morning and memantine 10 mg in the evening in Week 3; dose increase if tolerated to memantine 10 mg twice a day, in the morning and the evening Weeks 4 to 12.
Period: Overall Study
Arm/Group | Memantine | Placebo
Started | 48 | 24
Completed | 30 | 14
Not Completed | 18 | 10
Not completed — Lost to Follow-up | 6 | 3
Not completed — Lack of Efficacy | 5 | 3
Not completed — Adverse Event | 2 | 2
Not completed — Physician Decision | 1 | 0
Not completed — Withdrawal of consent | 4 | 2

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Memantine | Placebo | Total
Number analyzed (Participants) | 48 | 24 | 72
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.29 (10.48) | 47.33 (7.98) | 46.70 (9.54)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 11 | 35
  Male | 24 | 13 | 37
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 48 | 24 | 72

OUTCOME MEASURES:

1. Primary Outcome: California Verbal Learning Test (CVLT) at Week 12
Description: The CVLT is used to measure verbal learning and episodic long-term memory. It assesses learning, short- and long-delayed recall and recognition for a list of 16 shopping items. Subjects are expected to remember a list of words. They are asked to repeat the words remembered 5 times (5 trials). Each of the words correctly remembered, in each trial, is marked as 1 point. The reported data represent the number of correct items for the Trial 1, Trial 5, Short Delay Free Recall, and Long Delay Free Recall. The long-delayed recall is assessed at 20 minutes. The CVLT enables a comprehensive characterization of a participant's memory profile.
Time Frame: Week 12
Population: All Randomized participants with data available at Week 12.
Measure: Mean (Standard Deviation); unit: correct items
Arm/Group | Memantine | Placebo
Number analyzed (Participants) | 26 | 13
correct items
  CVLT Trial 1 | 11.88 (2.659) | 11.55 (2.505)
  CVLT Trial 5 | 11.63 (3.645) | 11.73 (3.524)
  CVLT Short Delay Free Recall | 11.79 (3.718) | 12.09 (3.477)
  CVLT Long Delay Free Recall | 14.46 (1.641) | 14.55 (1.128)

2. Primary Outcome: California Verbal Learning Test (CVLT) at Week 6
Description: as for outcome 1
Time Frame: Week 6
Population: All Randomized participants with data available at Week 6.
Measure: Mean (Standard Deviation); unit: correct items
Arm/Group | Memantine | Placebo
Number analyzed (Participants) | 41 | 19
correct items
  CVLT Trial 1 | 11.55 (3.280) | 10.65 (2.849)
  CVLT Trial 5 | 9.15 (3.815) | 9.05 (3.316)
  CVLT Short Delay Free Recall | 11.31 (4.335) | 10.24 (4.024)
  CVLT Long Delay Free Recall | 14.03 (2.732) | 13.53 (3.826)

3. Secondary Outcome: Rapid Visual Information Processing Task (RVP)
Description: RVP is a sensitive measure of sustained attention. In this test, a white box appears in the center of the screen with digits from 2-9 in a pseudorandom order at a rate of 100 digits per minute. Participants are asked to identify target sequences of three digits and to register responses using the press pad.
  RVPA is a measure of target sensitivity (i.e., the ability to discriminate between target and distractors). The outcome is defined as a z-score (statistical deviation from normal). A z-score of 0 is average. Higher z-scores represent better than average performance and negative z-scores represent worse than average performance.
  RVPB is an index of response bias (i.e., the tendency to respond or not respond in general). The outcome is defined as a z-score (statistical deviation from normal). A z-score of 0 is average. Higher z-scores represent a stronger tendency to respond and negative z-scores represent a less than average tendency to respond.
Time Frame: Weeks 6 and 12
Population: All randomized participants with data available at the given time-point.
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | Memantine | Placebo
Number analyzed (Participants) | 48 | 24
z-score
  RVPA, Week 6: number analyzed (Participants) | 41 | 19
  RVPA, Week 6 | -1.3997 (5.23534) | -0.6859 (0.96275)
  RVPA, Week 12: number analyzed (Participants) | 26 | 13
  RVPA, Week 12 | -0.1508 (1.49027) | -0.6017 (1.00486)
  RVPB, Week 6: number analyzed (Participants) | 41 | 19
  RVPB, Week 6 | -2.4440 (7.76338) | -0.2353 (0.74248)
  RVPB, Week 12: number analyzed (Participants) | 26 | 13
  RVPB, Week 12 | -1.4833 (4.39216) | -0.2108 (0.59609)

ADVERSE EVENTS:
Time Frame: 12 Weeks
Arm/Group | Memantine | Placebo
Serious Adverse Events (participants affected / at risk) | 0/48 | 0/24
Other Adverse Events (participants affected / at risk) | 0/48 | 2/24
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Memantine (N=48) | Placebo (N=24)
Gastric reflux (Gastrointestinal disorders) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No